CLINICAL TRIAL: NCT05804253
Title: Clinical, Radiographic and Histological/Histomorphometric Analysis of Maxillary Sinus Grafting With Deproteinized Porcine or Bovine Bone Mineral: a Randomized Controlled Clinical Trial
Brief Title: Maxillary Sinus Grafting With Deproteinized Porcine or Bovine Bone Mineral.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Camlog Oral Reconstruction Foundation (Other)
Responsible Party: Principal Investigator, Krennmair Gerald, Univ.Prof.Dr.Dr, Camlog Oral Reconstruction Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CamlogORF
Record Dates: First submitted 2023-03-14; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Histomorphometry
MeSH Terms: interventions — Sinus Floor Augmentation

STUDY DESIGN:
Intervention Model Description: randomized clinical trial.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bovine bone (Active Comparator): Patients received maxillary sinus augmentation grafting with bovine bone mineral
  Interventions: Procedure: Maxillary sinus augmentation
- Porcine bone mineral (Active Comparator): patients received maxillary sinus augmentation grafting with porcine bone mineral
  Interventions: Procedure: Maxillary sinus augmentation

INTERVENTIONS:
Procedure: Maxillary sinus augmentation — Maxillary sinus grafting with 2 different xenogenic materials

SUMMARY:
The present study aimed to compare the histomorphometrically evaluated new bone formation, the radiographically measured graft stability and the clinical implant outcome between maxillary sinuses grafted either with deproteinized porcine bone mineral (DPBM) or deproteinized bovine bone mineral (DBBM). Conclusions: From a clinical point of view, the present results demonstrate that DPBM provides for comparable bone formation and stable graft dimension and high implant success rates combined with healthy peri-implant condition:

DETAILED DESCRIPTION:
Materials and Methods: Thirty maxillary sinuses in 28 participants were initially included and randomly assigned to the test group (TG;DPBM: n=15) or the control group (CG,DBBM: n=15). After a healing period (6 months) bone core biopsies were axially retrieved in the molar site for histological/ histomorphometrical analysis of new bone formations. In addition, radiographically measured graft stability as well as the clinical implant outcome (implant survival/success/peri-implant health) were assessed at the 1-year and 3-year follow-up evaluations.

ELIGIBILITY:
Inclusion Criteria:

* maxillary sinus atrophy in the need of sinus augmentation, 2 stage augmentation procedure

Exclusion Criteria:

* drug abuse, additional augmentation procedure, heavy smokers, bisphosphonate abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
New bone formation | 3 year
  Bone trephine specimen retrieved at implant placement were histomorphometrically analyzed.
  With special interest % of new bone formation,% of residual graft and % of connective tissue were evaluated and compared between bovine and porcine mineral bone used for sinus grafting.

IPD SHARING:
Plan to Share IPD: No